CLINICAL TRIAL: NCT00199095
Title: Pilot Study for Treatment of Elderly Patients (>65 Years) With Acute Lymphoblastic Leukemia
Brief Title: Treatment of Elderly Patients (>65 Years) With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL11
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Elderly; Chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Doxorubicin; Cyclophosphamide; Cytarabine; Dexamethasone; Idarubicin; Ifosfamide; Methotrexate; Mercaptopurine; Teniposide; Vincristine

INTERVENTIONS:
Drug: Adriamycin
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Dexamethasone
Drug: Idarubicin
Drug: Ifosfamide
Drug: Methotrexate
Drug: Mercaptopurine
Drug: VM26
Drug: Vincristine

SUMMARY:
The aim of this study is to test feasibility and efficacy of a dose reduced chemotherapy in elderly patients with newly diagnosed acute lymphoblastic leukemia. The regimen consists of induction phase I and II followed by cyclic consolidation cycles, reinduction and maintenance therapy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute lymphoblastic leukemia (pro-B,common,pre-B,pre-T,Thy-,mature T, B-ALL)
* age > 65 years
* written informed consent
* Karnofsky > 50% (if not mainly caused by leukemia)
* laboratory at diagnosis or after supportive pre-treatment Creatinine < 2 mg/dl Uric Acid < 8 mg/dl Bilirubin < 1.5 mg/dl ALA, ASA,AP < 2.5 x ULN

Exclusion Criteria:

* severe second diseases (e.g. renal failure, cardiomyopathy etc., not caused by leukemia) that exclude treatment according to the protocol
* severe psychiatric illness or other circumstances which may compromise cooperation
* active second neoplasia
* clinical signs of life threatening infections or bleeding, uncontrollable prior to chemotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40
Dates: Start 1997-02 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Results of induction therapy,Distribution of entry criteria,Treatment feasibility,Relapse rate and localisation,Death in CR,Remission duration, survival and leukemia free survival,Prognostic factors,Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, Study Chair — University Hospital Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- See also: German Leukemia Trial Registry — http://www.studienregister-online.de